CLINICAL TRIAL: NCT01206192
Title: The Differential Effects of Intimate Terrorism and Situational Couple Violence on the Mental Health of Abused Chinese Women
Brief Title: Differential Effects of Intimate Partner Violence (IPV) on Mental Health
Status: Completed | Type: Observational
Sponsor: TIWARI, Agnes (Other)
Responsible Party: Sponsor-Investigator, TIWARI, Agnes, Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Other Study IDs: UW 10-095; GRF753510 (Other Grant/Funding Number: Research Grants Council Hong Kong)
Record Dates: First submitted 2010-09-19; First posted 2010-09-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Battered Women
Keywords: Intimate Terrorism; Situational couple violence; Mental health; Chinese; Women
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abused Chinese women

SUMMARY:
The purpose of this study is to extend the extant work on the typology of intimate partner violence (IPV) by employing mixed methods to collect quantitative and qualitative data.

DETAILED DESCRIPTION:
Although post-traumatic stress disorder and depression have been identified as the two most common consequences of intimate partner violence, research has generally not differentiated the effects of different types of intimate partner violence on victim's mental health. With intimate partner violence treated as a single phenomenon rather than having different types, abused women are unlikely to receive the most appropriate interventions.

Johnson's typology of control has been used increasingly to classify intimate partner violence based on physical assault and controlling behavior. Two distinct types of the violence, Intimate Terrorism and Situational Couple Violence, have received much attention. The two differ not only in the cause and trajectory of the violence but also in the effects including mental health outcomes. Although control is a critical factor in distinguishing intimate terrorism from situational couple violence, there is no consensus on what constitutes high or low control in physically violent intimate relationships. Partly, this may be due to the sole reliance on quantitative measures to determine the levels of control. By understanding the context in which control tactics are used, qualitatively different phenomena between violent relationships with high control and those with low control may be more apparent. Thus, there is a need to collect both quantitative and qualitative data on the use of controlling behaviors.

It has also been hypothesized that intimate terrorism and situational couple violence have different mental health outcomes but few studies have examined this empirically and none has studied women's experiences of the negative psychological consequences as victims of these two types of violence.

ELIGIBILITY:
Inclusion Criteria:

* Chinese women, aged 18 or above, from a shelter or a community centre, and screened positive for IPV in the past 12 months

Exclusion Criteria:

* Unable to communicate in Cantonese or Putonghua
* The perpetrator is not an intimate partner

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Shelter residents and community sample
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Intimate terrorism and situational couple violence among shelter and community-dwelling abused Chinese women | one-off

SECONDARY OUTCOMES:
Use of controlling behaviors | one-off
Post-traumatic stress disorder symptoms | one-off
Depression symptoms | one-off

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Tiwari, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Po Leung Kuk, Hong Kong, China

REFERENCES:
- [Derived] Tiwari A, Chan KL, Cheung DS, Fong DY, Yan EC, Tang DH. The differential effects of intimate terrorism and situational couple violence on mental health outcomes among abused Chinese women: a mixed-method study. BMC Public Health. 2015 Mar 31;15:314. doi: 10.1186/s12889-015-1649-x. PMID 25886388
- [Derived] Tiwari A, Cheung DS, Chan KL, Fong DY, Yan EC, Lam GL, Tang DH. Intimate partner sexual aggression against Chinese women: a mixed methods study. BMC Womens Health. 2014 May 25;14:70. doi: 10.1186/1472-6874-14-70. PMID 24886374